CLINICAL TRIAL: NCT00844987
Title: The Importance of Vascular Endothelial Growth Factor (VEGF), Hepatocyte Growth Factor (HGF) and Platelet Derived Growth Factor (PDGF) as a New Indicators of Myocardial Ischemic Injury in Comparison With Commonly Used Biomarkers.
Brief Title: Vascular Endothelial Growth Factor (VEGF), Platelet Derived Growth Factor (PDGF), Hepatocyte Growth Factor (HGF) in Patients With Acute Coronary Syndrome (ACS)
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Anna Konopka MD PhD, Institute of Cardiology, CCU, Warsaw, Poland
Other Study IDs: 2.32/II/06; 937
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Acute Coronary Syndrome
Keywords: PDGF; HGF; VEGF; ACS; markers of myocardial injury; Vascular Endothelial Growth Factor; Hepatocyte Growth Factor; Platelet Derived Growth Factor; Strategies in ACS
MeSH Terms: conditions — Acute Coronary Syndrome; Deafness, Autosomal Recessive 39

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The main aim of the study is a comparison of serum and plasma concentration of VEGF (Vascular Endothelial Growth Factor), HGF (Hepatocyte Growth Factor) and PDGF (Platelet Derived Growth Factor) with markers of myocardial injury as troponin I, hsCRP, CK-MB and NT-proBNP assessed in patients with first episode of acute coronary syndrome (ACS) in their lives and the estimation of assumed value of VEGF, HGF and PDGF in prognosis of cardiovascular complications at 3 months follow up especially with respect to myocardial infarction (MI), exacerbation of angina, reintervention (PTCA,CABG), symptoms of heart failure, stroke, rehospitalization due to cardiovascular reasons and death. The dynamics of changes in serum and plasma concentration of growth factors in comparison with values of myocardial injury markers will be checked. For the realization of the purpose of the study biochemical measurements will be performed twice i.e. just after admission to hospital and 24h later. Area of a myocardial injury will be estimated by echocardiography examination.

DETAILED DESCRIPTION:
In the recent years several biomarkers have been investigated to be used for diagnostic and risk stratification in patients with symptoms of acute coronary syndrome. Troponins are preferred markers for myocardial injury due to its high specificity and sensitivity what makes them superior than traditional cardiac enzymes as CK or CK-MB. Elevated level of NT-proBNP is a marker of heart failure strongly associated with increased mortality rate. This study is invented for searching new sensitive indicators of myocardial injury and predictors of bad outcome in patients with symptoms of ACS especially useful in difficult diagnostic and therapeutic situations.

The study is performed in patients with first episode of ACS in their life who are eligible for coronary angiography and eventually for PCI. All subjects who agree to participate in the study are informed of its nature and purpose. Patients, only due to the symptoms and according to ESC guidelines are referred for coronary angiography, primary PCI, surgery revascularisation and pharmacological treatment. Inclusion into the study does not influence on the type of the treatment. The measurements of VEGF, HGF, PDGF, troponin I, hsCRP, CK-MB and NT-proBNP are assessed twice i.e. as soon as possible after admission to hospital and 24h after the first measurements. For estimation of changes in concentration of growth factors in time in some patients the multiple assessments will be performed (9 measurements during first 24h and 1 before discharge from hospital). In healthy volunteers (10 to 20 subjects) one, control measurement of HGF will be performed. Three days after ACS symptoms appeared, left ventricular function is determined by echocardiography. Scheduled control visits are performed after 3 months follow up. The demographic and clinical data, duration of chest pain, results of 12 leads ECG, angiographic findings, haemodynamic description of cardiac function (parameters from echocardiography and ventriculography), type of invasive revascularisation and results of performed measurements and examinations will undergo single and multivariable statistical analysis. Additionally, according to a few clinical and angiographic findings for statistic analysis will be specified either:

subgroup of patients with "major myocardial injury" which will comprise patients with anterior or antero-lateral myocardial infarction (MI) with occlusion or significant left anterior descending (LAD) branch stenosis and/or multivessel disease,

subgroup of patients with "moderate myocardial injury" which will consist of patients with inferior and/or posterior MI and with singlevessel disease but not LAD,

subgroup of patients with "minor myocardial injury" which will include patients with NSTE-ACS (Non-ST-Segment Elevation ACS) and without a significant increase of myocardial injury markers.

ELIGIBILITY:
Inclusion Criteria:

1. typical chest pain;
2. ST segment elevation or depression in ECG;
3. indication for coronary angiography; if necessary with PCI and 4) signed inform consent.

Exclusion Criteria:

1. known past history of a myocardial infarction;
2. not signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Institute of Cardiology due to ACS
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Composite end point of the study which consists of: death, myocardial infarction, exacerbation of angina, heart failure, cardiovascular reintervention, rehospitalization due to cardiovascular reasons, stroke | 3 months

SECONDARY OUTCOMES:
Dynamics of serum and plasma concentration of VEGF, HGF and PDGF and comparison with changes of examined markers of myocardial injury and dysfunction | hospital stay
Left ventricular function | hospital stay
symptoms of heart failure | 3 months
symptoms of angina | 3 months
Death | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Konopka, PhD, Study Director — Institute of Cardiology, CCU
Locations (1):
- Institute of Cardiology, Coronary Care Unit, Warsaw, Poland

REFERENCES:
- [Derived] Konopka A, Janas J, Piotrowski W, Stepinska J. Hepatocyte growth factor - the earliest marker of myocardial injury in ST-segment elevation myocardial infarction. Kardiol Pol. 2013;71(8):827-31. doi: 10.5603/KP.2013.0194. PMID 24049022
- [Derived] Konopka A, Janas J, Piotrowski W, Stepinska J. Concentration of vascular endothelial growth factor in patients with acute coronary syndrome. Cytokine. 2013 Feb;61(2):664-9. doi: 10.1016/j.cyto.2012.12.001. Epub 2013 Jan 10. PMID 23313225
- [Derived] Konopka A, Janas J, Piotrowski W, Stepinska J. Hepatocyte growth factor--a new marker for prognosis in acute coronary syndrome. Growth Factors. 2010 Apr;28(2):75-81. doi: 10.3109/08977190903403984. PMID 19939200